CLINICAL TRIAL: NCT07011407
Title: Facial Recognition in Acute Illness - The FACIAL Study
Brief Title: The FACIAL Study Pilot
Status: Not yet recruiting | Type: Observational
Sponsor: Lancaster University (Other)
Collaborators: University of Central Lancashire (Other); East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Senior Lecturer in Integrative Physiology, Lancaster University
Other Study IDs: FHM-2024-4068-RECR-2
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adult
Keywords: Facial Characteristics; Exercise; Thermal Patterns; Facial Expression; Maximal Exercise Test
MeSH Terms: conditions — Motor Activity; Facial Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maximal Exercise Test — Healthy participants will be situated on a cycle ergometer fitted with a 12-lead ECG or chest-strap heart rate monitor. Data from the questionnaire will be stored in a study site file in a locked cabinet in an office. Baseline readings will be obtained whilst on the bike for 3 minutes before the subject embarks on a 3-minute warm-up at 50 Watts (W). The workload (watts) on the bike is then increased to a workload that corresponds to a heart rate of 120 bpm (gentle exercise). The workload will then be increased by 25-50W every three minutes until volitional exhaustion. Between each stage, there will be a 30s rest period where the participant will be cycling with minimal resistance ("freewheeling") but will be otherwise stationary on the cycle ergometer. Still images of the face and facial video recordings will be taken during a 30s rest period between increases in exercise intensity. A finger-prick blood sample (glucose & lactate) will be taken at the beginning and every 3 minutes.

SUMMARY:
Facial recognition is a non-invasive method for analysing facial characteristics and changes in facial expressions. There is evidence to suggest there may be a link between physiological health and facial expression patterns. Many medical conditions are associated with specific facial characteristics, with some related to inherited genetic conditions and others that have been acquired as a result of medical conditions such as stroke, nerve injuries and dementia. If successful, this technology could prove useful for studies evaluating the monitoring of acute or chronic illness. The proposed study will ask participants to do a maximal exercise test that will challenge the body, as a proof-of-principle, to see how this correlates with facial expressions. Depending on the study outcomes and future work, it could prove to be a useful tool and clinical application in healthcare for evaluating and tracking patient health and well-being. The investigators want to conduct a proof-of-principle study where physically stressed young and healthy participants (in the form of a maximal exercise test), whilst recording facial expressions, will be used to determine the relationship between physiological stress and changes in facial parameters.

DETAILED DESCRIPTION:
For this pilot study, no specific sample size calculation is required for this pilot study as this will recruit 15 participants for proof of concept. The outcomes from this research will lead to the identification of measurement parameters to be evaluated in future studies concerning facial characteristics and their parameters. This will inform the next steps in the application of the process to further healthy participants with the ultimate aim to translate this to research on a range of patient populations in elective and acute medical settings.

Video and still image capture will be undertaken using a camera mounted on a tripod in front of the participant whilst they are exercising. The data analysis mainly consists of four processing stages, including facial landmark detection, facial region identification, region-based facial analysis and data correlations, as illustrated in the diagram below. The facial landmark detection can label a total of 68 points in each face, which are in the predefined locations. Based on the facial landmark, the region identification can segment the face into different areas, such as brows, eyes, chin, etc. Then, the region-based analysis can be applied to facial data and extracts the geometry, colour, emotion and temperature information of the individual facial region and calculates their variations against time. Finally, vital sign reading and region-based facial data are analysed together by using statistical tools in order to identify their correlations and demonstrate how facial appearances change in different scenarios.

Lancaster University is the data owner/controller, and UCLAN will follow Lancaster's requirements of data management when the data is processed. The data will be transferred on an encrypted hard drive and stored on secure online storage by UCLAN data protection rules. The data will only be accessible to the FACIAL study collaborators and statisticians. Whilst sociodemographic and physiological data can be anonymised, the video recordings of facial expressions cannot. The two sets of data will be provided with separate research codes so that protected data cannot be linked to identities by anyone other than the study team. Processing of protected data such as ethnicity and biometric data is central to the research question and ultimately, might have efficacy in the treatment of high dependency patients in hospital care.

The FACIAL Study protocol has been formulated and reviewed by the FACIAL Steering Committee, and research will be carried out in line with the University of Central Lancashire and Lancaster University code of ethics. The FACIAL study will be carried out by the FACIAL steering committee as a collaboration between East Lancashire Hospitals NHS Trust, Lancaster University and the University of Central Lancashire.

The findings from this study will be presented at national or international conferences. Any facial images used for publication will be obtained with additional consent from the individuals. Manuscript(s) will be prepared for submission to a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35
* Male or female
* Capable of completing a maximal exercise test
* Answer "NO" to all variables in the Physical Activity Readiness questionnaire (PAR-Q)

Exclusion Criteria:

* Musculoskeletal injury
* Cardiovascular disease
* Neurological disease, stroke, or other disease that may affect facial expressions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants from the general public, inlcuding students and staff from the university.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in distance between facial features | 60 minutes
  Change in inter-feature distance (e.g., between eyes, mouth corners) during different phases of exercise, captured using video and still images to detect facial regions and landmarks. Unit: millimetres (mm).
Change in size and shape of facial features | 60 minutes
  Change in facial feature dimensions (e.g., width and height of eyes, mouth) and geometric shape indices during different phases of exercise. Additionally, captured using video and still images to detect facial regions and landmarks. Units: millimetres² or shape index (unitless).
Change in facial blood flow patterns | 60 minutes
  Regional blood flow variation across facial regions during exercise, captured through thermal imaging. Unit: perfusion units or arbitrary units (a.u.)
Change in facial temperature | 60 minutes
  Alterations in surface temperature across facial regions during exercise, measured with thermal imaging. Units: degrees Celsius (°C)
Change in facial skin colour | 60 minutes
  Variation in facial colour intensity and hue across regions during exercise, analysed from captured video, thermal imaging and still images. Unit of measure: RGB values

SECONDARY OUTCOMES:
Change in heart rate | 60 minutes
  Heart rate is recorded at rest, during exercise, and during recovery. Units: Beats per minute (bpm)
Change in heart rate variability (HRV) | 60 minutes
  Analysis of time and frequency domain HRV indices during different exercise stages. Units: Milliseconds (ms)
Change in blood glucose | 60 minutes
  Blood glucose levels are recorded at rest, during exercise, and recovery. Unit: millimoles per litre (mmol/L)
Change in Blood Lactate | 60 minutes
  Blood lactate recorded at rest, during exercise, and recovery. Units: millimoles per litre (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health and Medicine, Lancaster University, Lancaster, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This pilot study is a proof-of-principle study where we physically stress young, healthy participants (in the form of a maximal exercise test), whilst recording facial expressions, to determine the relationship between physiological stress and changes in facial parameters. The code developed from this pilot will be used as part of a PhD project at UCLan and is therefore novel. Individual participant data will not be shared externally at this time.